CLINICAL TRIAL: NCT00823160
Title: A Randomized Prospective Study of the Definitive Management of the Stable Haemopericardium Following Penetrating Cardiac Injury Utilising Subxyphoid Window and Drainage.
Brief Title: Surgical Management of Blood in the Pericardial Sac After Penetrating Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Associate Professor Andrew Nicol, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 266/2002
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2009-04

CONDITIONS: Heart Injuries
Keywords: Pericardial window; Sternotomy; Haemopericardium
MeSH Terms: conditions — Heart Injuries; Pericardial Effusion | interventions — Sternotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Sternotomy (Active Comparator): Patients who are randomized to a sternotomy after the finding of blood in the pericardial sac.
  Interventions: Procedure: Sternotomy
- 2: Subxyphoid window (Active Comparator): Patients who receive a subxyphoid window after the finding of blood in the pericardial sac.
  Interventions: Procedure: Subxyphoid window

INTERVENTIONS:
Procedure: Sternotomy — Sternotomy performed after finding blood in the pericardial sac
  Arms: 1: Sternotomy
Procedure: Subxyphoid window — Subxyphoid window performed after the finding of blood in the pericardial sac
  Arms: 2: Subxyphoid window

SUMMARY:
Penetrating wounds to the heart may present to the emergency unit with the presence of blood in the pericardial sac as determined on ultrasound. If these patients are stable, the study hypothesis is that they can be managed with a very simple surgical procedure called a subxyphoid pericardial window (SXW), in which the blood is drained from around the heart via a small skin incision below the rib cage. In all other centres in the world these cases are managed by open chest surgery called a sternotomy. The investigator's experience in dealing with these injuries is that this is unnecessary and requires a large amount of resources for no benefit to the patient.

In this study, patients are randomized to receive either open chest surgery (sternotomy) or the much smaller operation of the SXW. The patients are then followed up with respect to their hospital stay and any complications that they develop. Normally, a patient undergoing open chest surgery will stay in intensive care unit for a minimum of 2 days and have a total hospital stay of at least 7 days and be at risk of a number of complications such as pneumonia. Patients undergoing a SXW usually remain in hospital for a period of 3 days and do not require intensive care management.

The investigator's hypothesis is that in all these patients the heart injury has sealed and the patient is no longer in any danger. It is not necessary to perform open chest surgery on these patients.

DETAILED DESCRIPTION:
Introduction:

This will be the first prospective, randomized clinical study ever performed on penetrating cardiac injuries in the world literature. A group of patients with penetrating chest injuries will present haemodynamically stable, with blood in the pericardial sac diagnosed on ultrasound. The accepted international management of what is termed; "the stable haemopericardium" has been a median sternotomy. In our experience in Cape Town, when a median sternotomy is performed in these cases, any cardiac injury if present has already sealed or there is no cardiac injury. We feel that these patients should be managed with a much smaller and simpler operation that does not require admission to the intensive care unit post-operatively and this is merely drainage of the blood from around the pericardial sac via a subxyphoid window (SXW).

Method A SXW is performed under general anaesthetic and involves a 5 cm incision below the sternum. The pericardial sac can be opened and the blood drained. This small operation also allows the heart to be examined for any active bleeding. If there is active bleeding then obviously, a median sternotomy is required to fix the hole in the heart. If there is no active bleeding then the patient is randomized to either median sternotomy (the international norm) or the pericardial sac is merely drained with a soft drain and no further surgery is performed. The randomization is computer generated. The patients are documented with respect to intensive care stay and total hospital stay. Any complications are noted and the patients are then followed up in order to ensure that the patients who underwent the SXW alone are alive and well. This is essential to ensure the safety of this much smaller procedure for this condition. Informed consent is signed for each patient and all patients must be older than 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Haemodynamically stable
* Penetrating chest trauma
* Informed consent signed
* Over the age of 18 years
* Fully conscious

Exclusion Criteria:

* Known coagulopathy
* Traumatic septal defect
* Haemodynamically unstable
* No informed consent
* Decreased level of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2001-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
survival at discharge till 6-months post surgery. | from surgery till 6-months post operative.

SECONDARY OUTCOMES:
post-operative hospital stay | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Nicol, MD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Navsaria PH, Nicol AJ. Haemopericardium in stable patients after penetrating injury: is subxiphoid pericardial window and drainage enough? A prospective study. Injury. 2005 Jun;36(6):745-50. doi: 10.1016/j.injury.2004.08.005. Epub 2005 Mar 28. PMID 15910827
- [Derived] Nicol AJ, Navsaria PH, Hommes M, Ball CG, Edu S, Kahn D. Sternotomy or drainage for a hemopericardium after penetrating trauma: a randomized controlled trial. Ann Surg. 2014 Mar;259(3):438-42. doi: 10.1097/SLA.0b013e31829069a1. PMID 23604058